CLINICAL TRIAL: NCT05603663
Title: Genes and Health Behavior: the Impact of Awareness of High Polygenic Risk for Cardiovascular Disease on Health Behavior Among Young Overweight Adults
Brief Title: High Polygenic Risk and Health Behavior
Acronym: INTERVENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tartu (Other)
Collaborators: University of Helsinki (Other); The Estonian Health Insurance Fund (Unknown)
Responsible Party: Principal Investigator, Mikk JÜRISSON, Associate Professor of Public Health, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Grant #101016775
Record Dates: First submitted 2022-10-18; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Experimental): Young (25-44 years) overweight adults with high (top 20%) CVD PRS. The participants will be informed about their high PRS at the start of the study, calculated the overall CVD risk, and provided counseling and treatment of hypertension and/or high cholesterol if appropriate.
  Interventions: Genetic: Informing study subjects about their high CVD polygenic risk score
- Control group #1 (No Intervention): Young (25-44 years) overweight adults with high (top 20%) CVD PRS. The participants will be informed about the overall CVD risk and provided counseling and treatment of hypertension and/or high cholesterol if appropriate. The participants will be informed about their high PRS only at the end of the study.
- Control group #2 (No Intervention): Young (25-44 years) overweight adults with low (bottom 20%) CVD PRS. The participants will be informed about the overall CVD risk and provided counseling and treatment of hypertension and/or high cholesterol if appropriate. The participants will be informed about their low PRS only at the end of the study.

INTERVENTIONS:
Genetic: Informing study subjects about their high CVD polygenic risk score — During a visit, the family physician will announce the value of the subject's polygenic risk for CVD (either at the start or end of the trial, depending on the group) and discuss what it means, calculate the subject's overall risk for CVD using the Kardiokompass tool, advise the subject on weight loss and physical activity, and, if necessary, commence preventive treatment. Between visits, a mobile application will be utilized to collect data about the subjects' level of physical activity and body weight as well as to send reminders to the subjects every two weeks regarding exercise and healthy lifestyle choices.
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to evaluate the impact of awareness of high polygenic risk for CVD on health behavior among young overweight adults. We want to evaluate the impact of awareness of high polygenic risk for CVD on body mass index within 12 months, the impact of awareness of high polygenic risk for CVD on other health indicators (physical activity, systolic blood pressure, cholesterol and triglyceride levels, smoking, waist circumference, CVD risk score), and assess the cost-effectiveness of informing people about the high polygenic risk for CVD.

The trial will be conducted in a primary care setting, for which the high genetic-risk subjects will be invited to visit their family physician. In the course of the first visit, the family physician will assess the participant's health status and will counsel the participant on healthy choices for increasing their level of physical activity and losing weight. If necessary, the family physician will start treatment to lower the participant's blood pressure or cholesterol following current treatment guidelines. The participants in the intervention group will be informed of their high polygenic risk for CVD at the start of the study, while the control subjects at the end of the study. There will be three study visits at 6-month intervals. Between visits, the participants will receive reminders via a mobile health application to change their health behavior. At the end of the trial (month 12), the health indicators of the participants will be assessed and compared between the three trial groups. If a significant difference in BMI is found, it will presumably be related to the fact of learning of the high genetic risk, in which case the use of genetic data in primary prevention may be considered effective.

DETAILED DESCRIPTION:
Background

Cardiovascular disease (CVD) is the most prevalent cause of mortality. The risk of CVD can be reduced through effective prevention measures.

The risk of CVD can be assessed using genetic analysis. Large-scale international studies have shown that CVD is a polygenic disease. Based on the interaction of multiple single-nucleotide polymorphisms (SNPs) in individuals, a polygenic risk score (PRS) methodology has been developed for individual risk assessments.

Assessment of polygenic risk for CVD is not yet employed in clinical practice, as it is not clear whether awareness of high risk motivates health behavior to make healthier choices to prevent the related illness. Existing research results are contentious. For example, it is not clear whether informing smokers of their high genetic risk for cancer contributes to their quitting smoking or whether physical activity increases in individuals with a high PRS for diabetes after learning of their genetic risk. As the risk of disease in individuals with a high PRS can be reduced predominantly through healthy choices, knowledge of these issues is important for the inclusion of PRS in treatment guidelines.

Hypothesis

Learning of high polygenic risk changes people's health behavior, increasing the impact of personalized primary prevention of CVD.

Aim of the study

The primary objective of the trial is to evaluate the impact of awareness of high polygenic risk for CVD on health behavior among young overweight adults.

Objectives

1. To evaluate the impact of awareness of high polygenic risk for CVD on body mass index within 12 months (primary objective).
2. To evaluate the impact of awareness of high polygenic risk for CVD on other health indicators (physical activity, systolic blood pressure, cholesterol and triglyceride levels, smoking, waist circumference, and CVD risk score).
3. To evaluate the economic impact of informing people about the high polygenic risk for CVD.

Outcomes

1. Body mass index
2. Systolic blood pressure
3. Total cholesterol
4. Waist circumference
5. Smoking prevalence
6. Physical activity
7. CVD risk score

At the start and end of the trial, the participating physicians and family nurses will also be asked for their opinion on the utility of using data about genetic risk for CVD and genetic feedback (in the form of an anonymous survey).

Study design

To assess the health impacts of learning about the high polygenic risk for CVD, a randomized controlled trial will be conducted in a primary care setting, under real-life conditions.

The subjects will consist of 1500 individuals aged 25-44 years from the Biobank of the Estonian Genome Center (EGC) who are overweight and have no previously diagnosed CVD, and who belong to the top 20th percentile of polygenic risk for CVD (n=1000) and the bottom 20th percentile of polygenic risk for CVD (n=500). The high-PRS subjects will be randomized to two study groups, 500 in the intervention group and 500 in the 1st control group. The rest of the study subjects (500 subjects with low PRS) will be recruited for the 2nd control group from the Biobank database using matching for age and sex.

The trial will be conducted in a primary care setting, for which the high-PRS subjects from the intervention group and 1st control group will be invited to visit their family physician. In the course of the first visit, the family physician will assess the subject's health status and will counsel the subject on healthy choices for increasing their level of physical activity and losing weight. If necessary, the family physician will start treatment to lower the subject's blood pressure or cholesterol following current treatment guidelines. The subjects in the intervention group will be informed of their high polygenic risk for CVD by the family physician, while the control subjects will not be informed of the level of their polygenic risk. There will be three study visits at 6-month intervals. Between visits, the subjects will receive reminders to change their health behavior via a mobile application. At the end of the trial (month 12), the BMI, level of physical activity, and other health indicators of the subjects will be compared between the two trial groups. If a significant difference in BMI is found, it will presumably be related to the fact of learning of the high genetic risk, in which case the use of genetic data in primary prevention may be considered effective.

As the trial will assess the impact of awareness of high genetic risk, the physicians and controls must be completely blinded to their high genetic risk. To ensure the blinding of the family physicians, another control group (2nd control group, n=500) consisting of age- and sex-matched subjects with low CVD PRS are included in the trial. The genetic risk of the subjects in neither control group will be reported to the family physicians. Both control groups are mixed for family physicians. Thus, whenever a new control subject enters the trial, he/she may have either a high or low polygenic risk and the physician will not be able to distinguish between the two. This design ensures that the physicians are blinded to the risk of controls, and minimizes the risk of information bias.

The EGC will contact the selected gene donors based on the selection criteria by sending them a written invitation to participate in the study. In the invitation, the gene donors will be informed that the trial relates to personalized prevention of CVD and requires that the donor's health status parameters be assessed by a healthcare professional. The invitation will not contain any references to the extent of the individual's genetic risk. The initial consent will be sought for learning the polygenic risk score (PRS), for reporting the PRS to the subject's family physician, and for participating in the trial. Such consent ensures that the subjects are sufficiently informed to be able to participate in the study, while certain details of the trial, including the genetic risk, will only be disclosed to the subjects later by their family physician.

After having obtained the initial consent from the subjects the high-PRS subjects will be randomized and the low-PRS subjects matched to the intervention group. The EGC will thereafter transmit the study subjects' data (names, ID-s) to the family physicians. The PRS data will be extended for the intervention group subjects only. The PRS-s for controls will be extended at the end of the follow-up period. The family physicians will contact the subjects and schedule the first visit, during which they will present detailed information about the trial and obtain informed consent from participants. Blinding the controls will ensure that any changes in health behavior during the trial are not connected to the high PRS. At the end of the trial, the controls will be informed of their genetic risk and provided counseling and treatment similar to that for the intervention group at the first visit.

Sampling and power calculation

The sampling frame for the trial will consist of all of the EGC's gene donors (202,282 individuals as of 1 January 2022). The target group will be selected from the EGC's database from among gene donors who are not suffering from CVD or diabetes, based on their PRS, BMI, and age. The sample will consist of surviving males and females aged 25-44 who are overweight (BMI 25-29.99), belong to the top or bottom quintile for polygenic risk for CVD,m, and have not been diagnosed with CVD.

According to a preliminary query, the EGC's database contains data on about 2,000 individuals with a high PRS for CVD (top quintile) and about 2,000 individuals with a low PRS for CVD (bottom quintile) who are aged 25-44, have not been diagnosed with CVD and have a BMI of 25-29.99. 1300 of the approximately 2,000 individuals proven to belong to the highest quintile for polygenic risk for CVD will be selected for the intervention group and first control group of the trial, and approximately 650 of those in the lowest quintile for polygenic risk for CVD will be selected for the second control group, with the assumption of an average response rate of around 70% and a final number of subjects of up to 1,500 (500 in the intervention group, 1,000 in the control groups). The investigators calculated that the expected difference in the estimated 1-year BMI between the intervention (24 ±2.35) and control (23.6) groups should be detectable with a type 1 error of 0.05 and 1-the power of 0.20 with the total sample of >1000 high polygenic risk men and women from the Biobank database. To ensure the optimal number of physicians participating in the trial, the sampling will also be based on the practice lists of family physicians and will be conducted utilizing convenience sampling, by giving preference to practice lists that include larger numbers of subjects. Some of the family physicians who will be participating in the trial have already acted as partners to the EGC in the collection of the genetic data, which is also why their practice lists will likely include more subjects. The sampling will proceed from practice lists that include the greatest number of suitable gene donors to those with fewer potential subjects until the required number of subjects has been achieved.

Randomization

Randomization will involve the intervention group and the first control group. Randomization will be conducted at the EGC, as the family physicians will only be provided access to the data of the individuals on their practice list and the randomization cannot be carried out at their offices. The subjects in the second control group will be age- and sex-matched to the intervention group.

Intervention

The intervention consists of three activities:

1. Informing the participant about the polygenic risk and calculating the total disease risk. Only the intervention group participants will be informed about the high polygenic risk.
2. Health counseling
3. Initiating preventive treatment of high blood pressure and/or high cholesterol. During a visit, the family physician will announce the subject's polygenic risk for CVD (either at the start or end of the trial, depending on the group) and discuss what it means, calculate the subject's overall risk for CVD using the Kardiokompass tool, advise the subject on weight loss and physical activity, and, if necessary, commence preventive treatment. Between visits, a mobile application will be utilized to collect data about the subjects' level of physical activity and body weight as well as to send reminders to the subjects every two weeks regarding exercise and healthy lifestyle choices.

Treatment of subjects with high or moderate overall risk for CVD

Subjects with high or moderate overall risk will be advised on healthy lifestyle choices and, where necessary, provided preventive treatment by their family physician. All subjects will receive treatment according to the treatment guidelines of the European Society of Cardiology (ESC) and their personal risk score. Although this treatment of patients conforms to modern standard primary care practices, additional intervention guidelines will be drawn up in Estonian for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25-29.99
* High polygenic risk for cardiovascular disease confirmed
* Willing and able to participate in the trial
* Informed consent provided

Exclusion Criteria:

* Diagnosis of ischemic heart disease (I20-25)
* Diagnosis of stroke (I60-64, I69, G45)
* Diagnosis of peripheral vascular occlusion (I65-66, I67.2, I70, I73.9)
* Diagnosis of diabetes (E10-14)

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1540 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | 12 months
  The difference in mean BMI between study groups. Weight and height will be combined to report BMI in kg/m2

SECONDARY OUTCOMES:
Systolic blood pressure | 12 months
  The difference in mean systolic blood pressure in mm Hg between study groups
Total Cholesterol | 12 months
  The difference in mean total cholesterol between study groups. Total cholesterol is measured in mmol/l
Waist circumference | 12 months
  The difference between mean waist circumference in cm between study groups
Smoking prevalence | 12 months
  The difference between smoking prevalence between study groups. Smoking prevalence is calculated as a proportion of smokers in each study group
Physical activity | 12 months
  The difference between average weekly physical activity between study groups. The assessment of physical activity is based on estimated number of daily and weekly steps measured by mobile phone application and a validated self-assessment questionnaire SQUASH
Cardiovascular diseases 10-year risk | 12 months
  The difference in cardiovascular diseases 10-year risk between study groups. The risk assessment in disease probability in % is based on combination of age, sex, systolic blood pressure, total cholesterol, smoking status, and a polygenic risk score

CONTACTS AND LOCATIONS:
Overall Officials: Mikk JÜRISSON, PhD, Principal Investigator — University of Tartu
Locations (1):
- Institute of Family Medicine and Public Health, University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No